CLINICAL TRIAL: NCT02617485
Title: Randomized, Parallel-group, Double-blind, Comparative Bioequivalence Trial of MabionCD20 Compared to MabThera (Rituximab by Hoffman-La Roche) in Patients With Diffuse Large B-cell Lymphoma
Brief Title: MabionCD20 Compared to MabThera in Lymphoma Patients
Acronym: MADILYM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mabion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MabionCD20-002NHL
Record Dates: First submitted 2015-11-12; First posted 2015-12-01 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MabionCD20 (Experimental): A course of MabionCD20 consists of intravenous infusions in dose 375 mg/m2 body surface area, administered on day 1 of each chemotherapy cycle for 8 cycles.
  Intervention: Drug: Rituximab
  Interventions: Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: prednisone
- MabThera (Active Comparator): A course of MabThera consists of intravenous infusions in dose 375 mg/m2 body surface area, administered on day 1 of each chemotherapy cycle for 8 cycles.
  Intervention: Drug: Rituximab
  Interventions: Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: prednisone

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 IV on day 1 of each 21 days chemotherapy cycle. Number of Cycles: 8.
  Other Names: MabThera®, MabionCD20®
Drug: Doxorubicin — 50 mg of doxorubicin per square meter administrated IV on day 1 of each chemotherapy cycle
  Other Names: Hydroxydaunorubicin
Drug: Vincristine — 1.4 mg of vincristine per square meter, up to a maximal dose of 2 mg, administrated IV on day 1 of each chemotherapy cycle
  Other Names: Oncovine
Drug: Cyclophosphamide — 750 mg of cyclophosphamide per square meter of body-surface area administrated IV on day 1 of each chemotherapy cycle
Drug: prednisone — 100 mg of prednisone administrated PO per day for five days, day 1-5 of each chemotherapy cycle

SUMMARY:
The aim of the study is to demonstrate the high level of biosimilarity between MabionCD20 (MABION SA) and the reference product: MabThera (rituximab by Hoffman-La Roche) in patients with CD20-positive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Patients who meet criteria for participation in this study receive 8 intravenous infusions of MabionCD20® or MabThera® 21 days interval in combination with standard dosage regimen of CHOP. The duration of the study is 12 months. The treatment and observation period will last 26 weeks starting from Day 1, until Week 26 - one month after last IMP infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmed CD20 (cluster of differentiation 20) positive diffuse large B cell lymphoma (DLBCL)
2. Patients that had been diagnosed according to the WHO classification;
3. Performance status ≤ 2 on the ECOG (Eastern Cooperative Oncology Group) / WHO (world Health Organization) scale, performance status of 3 will be accepted if impairment is caused by DLBCL complications and improvement is expected once therapy is initiated;

Exclusion Criteria:

1. Life expectance less than 6 months;
2. Any chemotherapy, radiotherapy, immunotherapy, biologic, investigational or hormonal therapy for treatment of lymphoma within 28 days prior to treatment;
3. Rituximab, other anti-CD20 mAb (Monoclonal Antibodies) drug treatment, treatment with any cell depleting therapies - e.g., anti-CD4 (cluster of differentiation 4) anti-CD5 (cluster of differentiation 5), anti-CD3 (cluster of differentiation 3), anti-CD19 (cluster of differentiation 19), anti CD11 (cluster of differentiation 11), anti-CD22 (cluster of differentiation 11), BLys/BAFF (B Lymphocyte Stimulator/B-cell activating factor) within 1,5 years before screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- Bosnia and Herzegovina (4):
  - University Clinical Center Banja Luka, Banja Luka
  - University Clinical Center Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
  - General Hospital Zenica, Zenica
- Croatia (3):
  - GH "dr.Josip Bencevic", Slavonski Brod
  - CH Merkur, Zagreb
  - CHC Zagreb, Zagreb
- Georgia (3):
  - HEMA, Tbilisi
  - S. Khechinashvili state University clinic, Tbilisi
  - Medulla - Chemotherapy and Immunotherapy Clinic, Tbilisi
- Institut of Oncology, Hematology Department, Chisinau, Moldova
- Poland (4):
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Oddział Hematologiczny, Legnica
  - Samodzielny Publiczny Szpital Kliniczny nr1, Klinika Hematologii i Transplantacji Szpiku, Lublin
  - Szpital Wojewódzki w Opolu, Oddział Hematologii i Onkologii Hematologicznej, Opole
  - MTZ Clinical Research Sp. Z o.o., Warsaw
- Serbia (3):
  - Clinical Hospital Center Zemun, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Military Hospital Academy, Belgrade
- Ukraine (17):
  - Public utility "Chernivtsi regional clinical oncology dispensary", Day patient department, Chernivtsi
  - Municipal Institution "Dnipropetrovsk City multi-field Clinical Hospital #4", Oncology and medical radiology department, Dnipropetrovsk
  - Regional Clinical Hospital of Ivano-Frankivsk, Hematology Department., Ivano-Frankivsk
  - Regional Clinical Oncology Dispensary, Chemotherapy Department, Ivano-Frankivsk
  - Kharkiv Regional Clinical Oncology Centre, Deartment of haematology, Kharkiv
  - National Institute of Cancer, Department of chemotherapy, Kiev
  - Kiev City Clinical Oncological Center, Department of chemotherapy #2, Kiev
  - Utility Enterprise "Kirovograd regional oncology dispensary", Kirovohrad
  - Kryvyi Rih Oncology Dispensary, Dnipropetrovsk Highway, Kryvyi Rih
  - Volyn' Regional clinical hospital, Haematology Department, Lutsk
  - State institution "Institute for haemotopathology and haemotransfusion of National Academy of science of Ukraine, Lviv
  - Mykolayiv Region Clinical Hospital, Heamotology department, Mykolayiv
  - Poltava regional oncology hospital, heamotherapy department, Poltava
  - Regional clinical Hospital named after Novak, Hematology Department, Uzhhorod
  - Vinnitsya Regional Clinical Oncology Dispensary, Chemotherapy Department,, Vinnitsya
  - Regional Oncology dispensary, Zaporizhzhia
  - Zaporizhzhya Regional Clinical Hospital, Deartment of haematology and intensive therapy, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was initiated in 7 countries (Croatia, Bosnia and Herzegovina, Georgia, Moldova, Poland, Serbia, and Ukraine), but finally only 5 countries with 21 study sites recruited patients (Bosnia and Herzegovina, Georgia, Moldova, Poland, and Ukraine).
  Start date of recruitment: 29.03.2016
Pre-assignment Details: Screening lasted 28 days (from Day -35 to -8 before randomization), during which the eligibility status of patients was verified.
  Forty-eight patients were excluded before randomization: 45 patients did not meet eligibility criteria, one patient declined participation and two patients could not be randomized because of the limited availability of investigational drugs.
Groups:
- MabionCD20: Patients assigned to this arm received 375 mg/m2 of MabionCD20 intravenously every 3 weeks for 8 cycles on Days 1, 22 (Week 4), 43 (Week 7), 64 (Week 10), 85 (Week 13), 106 (Week 16), 127 (Week 19), and 148 (Week 22).
  Patients randomly assigned to MabionCD20 were followed up until Week 46.
- MabThera: Patients assigned to this arm received 375 mg/m2 of MabThera intravenously every 3 weeks for 8 cycles on Days 1, 22 (Week 4), 43 (Week 7), 64 (Week 10), 85 (Week 13), 106 (Week 16), 127 (Week 19), and 148 (Week 22).
  Patients randomly assigned to MabThera were followed up until Week 46.
Period: Treatment and Observation Period
Arm/Group | MabionCD20 | MabThera
Started | 100 | 40
Completed | 85 | 35
Not Completed | 15 | 5
Not completed — Adverse Event | 9 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Patient needed radiotherapy | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Physician Decision | 0 | 1
Period: Follow-up Period
Arm/Group | MabionCD20 | MabThera
Started | 85 | 35
Completed | 70 | 29
Not Completed | 15 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 2 | 1
Not completed — Need for CNS prophylaxis | 1 | 0
Not completed — Patient needed radiotherapy | 9 | 5
Not completed — Patient needed bone marrow transplantation | 1 | 0

BASELINE CHARACTERISTICS:
Population: SAF (all patients randomized into the study and receiving at least one infusion of MabionCD20 or MabThera).
Groups:
- MabionCD20: Patients assigned to this arm received 375 mg/m2 of MabionCD20 intravenously every 3 weeks for 8 cycles on Days 1, 22 (Week 4), 43 (Week 7), 64 (Week 10), 85 (Week 13), 106 (Week 16), 127 (Week 19), and 148 (Week 22).
- MabThera: Patients assigned to this arm received 375 mg/m2 of MabThera intravenously every 3 weeks for 8 cycles on Days 1, 22 (Week 4), 43 (Week 7), 64 (Week 10), 85 (Week 13), 106 (Week 16), 127 (Week 19), and 148 (Week 22).
- Total: Total of all reporting groups
Arm/Group | MabionCD20 | MabThera | Total
Number analyzed (Participants) | 100 | 40 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 29 | 107
  >=65 years | 22 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.2) | 54.3 (13.5) | 52.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 20 | 74
  Male | 46 | 20 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 100 | 40 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BSA [Mean (Standard Deviation); unit: cubic metre] | 1.9 (0.2) | 1.8 (0.2) | 1.8 (0.2)
Body weight [Mean (Standard Deviation); unit: kilograms] | 76.2 (17.4) | 73.6 (17) | 75.5 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From Day 1 to Week 4 (AUC[1-4])
Description: Area under the serum concentration-time curve from time zero (Day 1) to final time point measured after the first administration (Week 1) until Week 4 (AUC(W1-W4)). PK blood samples for this endpoint were drawn at Day 1 (before and after the first infusion), Day 8 ± 1 (7 days after first infusion), Day 15 ± 1 (14 days after first infusion), Day 22 ± 2 (before and after completion of the second infusion).
Time Frame: Baseline to Week 4
Population: PP W1-4 set (subset of ITT population based on patients without major protocol deviations to Week 4 (visit 4) and having a PK assessment on this visit. Completion of the study was not necessary for inclusion into this population).
Measure: Mean (Standard Deviation); unit: (μg*day)/mL
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 94 | 35
(μg*day)/mL | 1559.51 (358.092) | 1509.79 (382.559)
Statistical Analysis 1: Comparison: MabionCD20 vs MabThera; Estimated Geo LS-means ratio; Test type: Equivalence — Equivalence met if the 90% CI of the Geo LS Means ratio is contained with the pre-specified equivalence margin of 70% - 143%; Ratio of Geo LS-means = 1.0406, 90% CI 2-sided [0.9565 to 1.1321]

2. Primary Outcome: Area Under the Serum Concentration-time Curve From Week 13 to Week 26 (AUC[W13-W26])
Description: Area under the serum concentration-time curve from time zero to final time point measured from Week 13 until Week 26 (AUC[W13-W26]). PK blood samples for this endpoint were drawn at Day 85 ± 4 (before and after completion of the fifth infusion), Day 106 ± 4 (before and after completion of sixth infusion), Day 127 ± 4 (before and after completion of the seventh infusion), Day 148 ± 4 (before and after completion of the eight infusion), Day 155 ± 4 (one week after last infusion) and Day 176 ± 4 (one month after last infusion).
Time Frame: Week 13 to Week 26
Population: PP W13-26 set (subset of ITT population based on patients without major protocol deviations and having a PK assessment from Week 13 to Week 26).
Measure: Mean (Standard Deviation); unit: (μg*day)/mL
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
(μg*day)/mL | 16498.9 (3492.39) | 15647.4 (3629.83)
Statistical Analysis 1: Comparison: MabionCD20 vs MabThera; Estimated Geo LS-means ratio; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geo LS-means = 1.0611, 90% CI 2-sided [0.9822 to 1.1464]

3. Secondary Outcome: Ctrough (Before 8th Infusion)
Description: Trough serum concentration measured at the end of a dosing interval at steady state, taken directly before eighth infusion.
Time Frame: Week 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
μg/mL | 102.246 (43.897) | 90.61 (41.994)

4. Secondary Outcome: Cmax (Post 5th and 8th Infusion)
Description: Maximum serum drug concentration (Cmax) at steady state after the 5th and 8th infusions.
Time Frame: Week 13 (5th infusion) and Week 22 (8th infusion)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
μg/mL
  5th infusion | 273.356 (65.452) | 266.439 (66.086)
  8th infusion | 296.784 (58.295) | 296.462 (69.641)

5. Secondary Outcome: Kel (Post 5th and 8th Infusions)
Description: Elimination Rate Constant at steady stade after the 5th and 8th infusions.
Time Frame: Week 13 (5th infusion) and Week 22 (8th infusion)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
1/day
  5th infusion | 0.05663 (0.01794) | 0.05418 (0.01884)
  8th infusion | 0.04335 (0.01528) | 0.04379 (0.0123)

6. Secondary Outcome: T1/2 (Post 5th and 8th Infusions)
Description: Elimination half-life at steady state after the 5th and 8th infusions.
Time Frame: Week 13 to Week 16 and Week 22 to Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
days
  5th infusion | 14.801 (12.218) | 15.217 (7.889)
  8th infusion | 18.301 (7.92) | 16.997 (4.515)

7. Secondary Outcome: CLss (Post 5th and 8th Infusions)
Description: Clearance at steady state after the 5th and 8th infusions.
Time Frame: Week 13 to Week 16 and Week 22 to Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 74 | 29
mL/day
  5th infusion | 198.701 (53.427) | 206.905 (78.213)
  8th infusion | 179.168 (58.509) | 191.272 (89.016)

8. Secondary Outcome: AUC (W1-W26) B-cell
Description: Area under the serum concentration-time curve of CD19+ B cell counts, measured from the first administration to the final time point at Week 26 (AUC(1-26) B-cell).
Time Frame: baseline to Week 26
Population: ITT set (a subset of safety population based on patients who had at least one complete post baseline assessment of the area under the serum concentration-time curve from time zero to final time point (AUC(0-t)), measured after the first administration (Week 1) until the second administration at Week 4(AUC(1-4)).
Measure: Mean (Standard Deviation); unit: cells*days/mL blood
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 98 | 38
cells*days/mL blood | 3395.82 (22364.5) | 10476.2 (56943.0)

9. Secondary Outcome: AUC (W1-W26)
Description: Area under the serum concentration-time curve measured after the first administration (Week 1) until Week 26 (AUC(1-26))
Time Frame: Week 1 until Week 26
Population: PP W1-W26 set
Measure: Mean (Standard Deviation); unit: (μg*day)/mL
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 71 | 28
(μg*day)/mL | 28413.6 (5194.98) | 26955.3 (5849.22)

10. Secondary Outcome: Efficacy Assessment at Week 26
Description: An efficacy assessment was made after 8 treatment cycles (at Week 26) based on tumour responses classified according to the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas (Cheson et al. 1999). Response was assessed based on clinical, radiologic (CT scan) and pathologic (bone marrow) criteria. Possible efficacy responses were: complete response, partial response, stable disease, and progressive disease. Efficacy reported here includes all patients included in the ITT set.
Time Frame: Week 26
Population: ITT population including all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 100 | 40
Participants
  Complete | 34 | 14
  Partial | 42 | 18
  Stable disease | 10 | 4
  Progressive disease | 10 | 2
  Missing | 4 | 2

11. Secondary Outcome: Adverse Events
Description: Percentage of patients with at least one AE in a given category. Data from the entire follow-up are included (Period 1 and Period 2).
Time Frame: from baseline to Week 46
Population: SAF set (all patients randomized into the study and receiving at least one infusion of MabionCD20 or MabThera).
Measure: Number; unit: percent
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 100 | 40
percent
  all AEs | 71.0 | 67.5
  TEAEs | 71.0 | 65.0
  TESAEs | 19.0 | 12.5
  severe TEAEs | 40.0 | 22.5
  related TEAEs | 53.0 | 42.5
  related severe TEAEs | 29.0 | 22.5
  related TESAEs | 13.0 | 5.0
  TEAEs leading to death | 8.0 | 0
  related TEAEs leading to death | 2.0 | 0

12. Other Pre Specified Outcome: Immunogenicity
Description: Percentage of patients with positive ADA or NAb results in a given category. Data pertain to the entire follow-up period (from Baseline to Week 46).
Time Frame: from baseline to Week 46
Population: SAF set (sample from one patient not collected)
Measure: Number; unit: participants
Arm/Group | MabionCD20 | MabThera
Number analyzed (Participants) | 99 | 40
participants
  Treatment-induced ADA | 6 | 1
  Persistent ADA | 4 | 1
  Transient ADA | 2 | 0
  Treatment-boosted ADA | 0 | 0
  NAb positive | 0 | 0

ADVERSE EVENTS:
Time Frame: 46 weeks
Description: AEs were collected at each trial visit and followed up 30 days after patients completed the trial.
Arm/Group | MabionCD20 | MabThera
All-Cause Mortality (participants affected / at risk) | 8/100 | 0/40
Serious Adverse Events (participants affected / at risk) | 19/100 | 5/40
Other Adverse Events (participants affected / at risk) | 70/100 | 26/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MabionCD20 (N=100) | MabThera (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MabionCD20 (N=100) | MabThera (N=40)
Anaemia (Blood and lymphatic system disorders) | 14 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 22 | 10
Neutropenia (Blood and lymphatic system disorders) | 29 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 1
Hyperthermia (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 0
Respiratory tract infection (Infections and infestations) | 7 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminitransferase increased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 8 | 4
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 3 | 2
White blood count decreased (Investigations) | 9 | 4
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 5
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02617485/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT02617485/SAP_001.pdf